CLINICAL TRIAL: NCT07085949
Title: Evaluation of the Effect of Different Positive End-Expiratory Pressure (PEEP) Levels on Optic Nerve Sheath Diameter in Patients Undergoing Vertebral Surgery; Prospective Observational Study
Brief Title: Effect of Different Positive End-Expiratory Pressure (PEEP) Levels on Optic Nerve Sheath Diameter
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Karaşah Yalçın, MD, Izmir City Hospital
Other Study IDs: OPTIC NERVE
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: PEEP; Optic nerve sheath diameter; Intracranial Pressure Increase; spinal surgery
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEEP 5: 5 cmH2O PEEP will be administered during mechanical ventilation
  Interventions: Other: 5 cmH2O PEEP
- PEEP 10: 10 cmH2O PEEP will be administered during mechanical ventilation
  Interventions: Other: 10 cmH2O PEEP

INTERVENTIONS:
Other: 5 cmH2O PEEP — 5 cmH2O PEEP will be administered during mechanical ventilation
  Groups: PEEP 5
Other: 10 cmH2O PEEP — 10 cmH2O PEEP will be administered during mechanical ventilation
  Groups: PEEP 10

SUMMARY:
The goal of this prospective observational study is to evaluate the effects of different PEEP values on the optic nerve sheath diameter (ONSD), a noninvasive indicator of intracranial pressure (ICP), in patients undergoing vertebral surgery. The main question it aims to answer is how mechanical ventilation setting of 5 and 10 cmH2O PEEP effect optic nerve sheath diameter after surgery at extubation.

DETAILED DESCRIPTION:
During general anesthesia, endotracheal intubation can cause varying degrees of alveolar collapse, particularly in the lower lung regions, in 15-20% of cases. Postoperative atelectasis and pulmonary infections are responsible for both prolonged hospital stays and increased mortality and morbidity. Positive end-expiratory pressure (PEEP) combined with low tidal volume, defined as lung-protective ventilation strategies, is used in anesthesia practice because it prevents pulmonary barotrauma, improves pulmonary function, and reduces postoperative pulmonary complications. PEEP can prevent atelectasis and reduce the risk of ventilator-associated lung injury. PEEP at 10 cmH2O or less can be used without causing a significant increase in intracranial pressure or a significant decrease in cerebral perfusion pressure.

For years, low PEEP was used in neurosurgery and neurosurgical intensive care patients, considering that PEEP could increase ICP. However, recent studies in normovolemic patients without hypotension have shown that even with increased PEEP, no clinically significant increase in ICP was observed.

The optic nerve is anatomically an extension of the central nervous system. Cerebrospinal fluid (CSF) circulates within this extension, which is surrounded by dura mater. Therefore, noninvasive ultrasonographic measurement of optic nerve sheath diameter (ONSD) has been shown to be effective in detecting increased intracranial pressure (ICP) due to the reflection of changes in subarachnoid space pressure and CSF on the optic nerve sheath. An optic nerve sheath diameter greater than 6 mm is a noninvasive indicator of increased intracranial pressure.

The effect of positive end-expiratory pressure (PEEP) on optic nerve sheath diameter in patients undergoing vertebral surgery will be evaluated.

Optic nerve sheath diameter measurements will be taken twice with ultrasound, once before surgery in the preoperative waiting room and once after surgery in the postoperative recovery unit.

Hemodynamic data (systolic blood pressure, diastolic blood pressure, mean blood pressure, heart rate, peripheral oxygen saturation), and PEEP values during anesthesia will be recorded on the anesthesia observation form.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* ASA I, II, III
* Patients undergoing elective vertebral surgery in the prone position

Exclusion Criteria:

* Patients were defined as having a hemoglobin concentration below 9 g/dL
* Congestive heart failure
* Uncontrolled hypertension
* Severe COPD
* Pulmonary edema
* Cerebrovascular disease
* Those who have had carotid stenosis or surgery
* Hemodynamic instability
* Pregnant women
* Those who did not wish to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter measurement after extubation | just after extubation
  optic nerve sheath diameter will be measured at the end of the surgery after extubation

SECONDARY OUTCOMES:
heart rate0 | pre-induction
heartrate1 | up to 5 minutes after anesthesia induction
heartrate2 | up to 10 minutes after anesthesia induction
heartrate3 | up to 15 minutes after anesthesia induction
heartrate4 | up to 5 minutes after prone position
heartrate5 | up to 10 minutes after prone position
heartrate6 | up to 15 minutes after prone position
heartrate7 | up to 30 minutes after prone position
heartrate8 | up to 1 hour after prone position
heartrate9 | up to 2 hour after prone position
heartrate10 | up to 3 hour after prone position
mean arterial pressures0 | pre induction
mean arterial pressures1 | up to 5 minutes after anesthesia
mean arterial pressures2 | up to 10 minutes after anesthesia induction
mean arterial pressures3 | up to 15 minutes after anesthesia induction
mean arterial pressures4 | up to 5 minutes after prone position
mean arterial pressures5 | up to 10 minutes after prone position
mean arterial pressures6 | up to 15 minutes after prone position
meanarterialpressures7 | up to 30 minutes after prone position
meanarterialpressures8 | up to 1 hour after prone position
meanarterialpressures9 | 2 hour after prone position
meanarterialpressures10 | 3 hour after prone position
diastolicpressures0 | pre induction
diastolicpressures1 | up to 5 minutes after anesthesia induction
diastolicpressures2 | up to 10 minutes after anesthesia indüction
diastolicpressures3 | up to 15 minutes after anesthesia induction
diastolicpressures4 | up to 5 minutes after prone position
diastolicpressures5 | up to 10 minutes after prone position
diastolicpressures6 | up to 15 minutes after prone position
diastolicpressures7 | up to 30 minutes after prone position
diastolicpressures8 | up to 1 hour after prone position
diastolicpressures9 | up to 2 hour after prone position
diastolicpressures10 | up to 3 hour after prone position
systolicpressures0 | pre-induction
systolicpressure1 | up to 5 minutes after anesthesia
systolicpressure2 | up to 10 minutes after anesthesia
systolicpressure3 | up to 15 minutes after anesthesia
systolicpressure4 | up to 5 minutes after prone position
systolicpressure5 | up to 10 minutes after prone position
systolicpressure6 | up to 15 minutes after prone position
systolicpressure7 | up to 30 minutes after prone position
systolicpressure8 | up to 1 hour after prone position
systolicpressure9 | up to 2 hour after prone position
systolicpressure10 | up to 3 hour after prone position
peripheral oxygen saturation (SpO₂)0 | pre-ınduction
peripheral oxygen saturation (SpO₂)1 | up to 5 minutes after anesthesia induction
peripheral oxygen saturation (SpO₂)2 | up to 10 minutes after anesthesia induction
peripheral oxygen saturation (SpO₂)3 | up to 15 minutes after anesthesia induction
peripheral oxygen saturation (SpO₂)4 | up to 5 minutes after prone position
peripheral oxygen saturation (SpO₂)5 | up to 10 minutes after prone position
peripheral oxygen saturation (SpO₂)6 | up to 15 minutes after prone position
peripheral oxygen saturation (SpO₂)7 | up to 30 minutes after prone position
peripheral oxygen saturation (SpO₂)8 | up to 1 hour after prone position
peripheral oxygen saturation (SpO₂)9 | up to 2 hour after prone position
peripheral oxygen saturation (SpO₂)10 | up to 3 hour after prone position

CONTACTS AND LOCATIONS:
Overall Officials: Zeki Tuncel Tekgül, Professor, Study Chair — Izmir City Hospital